CLINICAL TRIAL: NCT00727961
Title: Obligatory Post-Registration Open-Label, Non-Comparative Multicenter Study of Efficacy and Tolerance Rate of Caelyx as Monotherapy in Patients With Epithelial Ovarian Cancer, Resistant to Previous Platinum Therapy.
Brief Title: A Study to Evaluate Efficacy and Tolerance of Caelyx in Patients With Epithelial Ovarian Cancer. (Study P04072)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04072
Record Dates: First submitted 2008-06-23; First posted 2008-08-05 (Estimated); Results first posted 2009-07-16 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Caelyx Intravenous, 50 mg/m^2, given for 6 cycles
  Interventions: Drug: Pegylated Liposomal Doxorubicin hydrochloride

INTERVENTIONS:
Drug: Pegylated Liposomal Doxorubicin hydrochloride — Caelyx Intravenous, 50 mg/m^2 (60 minute infusion) on day 1, every 4 weeks, during 6 cycles
  Other Names: Caelyx

SUMMARY:
The aim of this study is to evaluate efficacy and tolerability, and number of positive response to treatment with CAELYX (50 mg/m^2), administered as monotherapy once per 4 weeks to patients with metastatic epithelial ovarian cancer, resistant to previous platinum therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent and/or parent or legal guardian must have signed a written informed consent.
* Women must be greater than or equal to 18 years of age, of any race.
* Women of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active) must be using an acceptable method of birth control (e.g., hormonal contraceptive, medically prescribed IUD, condom in combination with spermicide) or be surgically sterilized (e.g., hysterectomy or tubal ligation).
* Morphology (cytology or histology) confirmed diagnosis of epithelial ovarian cancer.
* Patients with 1 or more measurable and/or evaluable tumors, according to the results of CT, MRT scans or X-ray, etc.
* Patients, including those after primary surgical treatment, who had previously received platinum chemotherapy and in whom second-line therapy is indicated.
* Karnofsky performance status above 60%.
* Left ventricular ejection fraction above 50% (according to the results of echocardiography).
* Adequate bone marrow function as indicated by:

  * Platelets >100x10^9/L
  * Haemoglobin > 9 g/dL
  * Absolute neutrophil count >1.5x10^9/L
* Adequate renal function as indicated by:

  * Serum creatinine < 1.5 х ULN
* Adequate liver function as indicated by:

  * Bilirubin level and AST or ALT activity < 2 х ULN (with the exception of cases related to primary disease).

Exclusion Criteria:

* Women who are pregnant or nursing.
* Subjects who have not observed the designated washout periods for any of the prohibited medications.
* Subjects who have used any investigational product within 30 days prior to enrollment.
* Medical history indicating serious concomitant diseases, such as congestive heart failure of II NYHA class or higher, insulin-dependent diabetes mellitus, clinically significant liver disease, mental disorders.
* Non-controlled bacterial, viral or fungal infections.
* Conditions and reasons (medical, social and psychological) that might prevent adequate follow-up of patients.
* Any other active primary tumor under treatment (except basal or squamous cell carcinoma or in situ cervix carcinoma).
* Patient has symptomatic metastasis to brain.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2004-11-09 (Actual); Primary Completion 2008-01-10 (Actual); Study Completion 2008-01-10 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Caelyx Intravenous: Caelyx Intravenous, 50 mg/m^2, given for 6 cycles
Period: Overall Study
Arm/Group | Caelyx Intravenous
Started | 58
Completed | 21
Not Completed | 37
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 4
Not completed — Patient's refusal | 2
Not completed — Progression | 30

BASELINE CHARACTERISTICS:
Arm/Group | Caelyx Intravenous
Number analyzed (Participants) | 58
Age, Customized [Number; unit: participants] | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response
Description: Complete response was defined as complete disappearance of all measurable and assessable disease with no new disease or disease-related symptoms as measured by chest x-ray, computed tomography scan, and magnetic resonance imaging.
Time Frame: 4 weeks after chemotherapy completed
Measure: Number; unit: participants
Arm/Group | Caelyx Intravenous
Number analyzed (Participants) | 58
participants | 0

2. Secondary Outcome: Mean Time to Positive (Partial) Treatment Response Achievement
Description: Time to the occurence of partial effect achievement as measured by chest x-ray, computed tomography scan, and magnetic resonance imaging.
  Partial response required a 50 percent or greater decrease in the sum of the products of all bidimensionally measurable lesions without progression of any assessable disease and no new lesions.
Time Frame: from the beginning of study drug administration up to 4 weeks after chemotherapy completed
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Caelyx Intravenous
Number analyzed (Participants) | 58
days | 128.0000 (50.26430)

3. Secondary Outcome: Median Time to Progression
Description: Median time to the occurence of progression. Progression was defined as 25 percent or greater increase size of measurable lesion. Reappearance of lesion, worsening of assessable disease or appearance new lesions were considered progression as measured by chest x-ray, computed tomography scan, and magnetic resonance imaging.
Time Frame: from the beginning of study drug administration up to 4 weeks after chemotherapy completed
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Caelyx Intravenous
Number analyzed (Participants) | 58
days | 98.0 [88.8 to 107.2]

4. Secondary Outcome: Mean Survival Time During the Study
Description: Mean time to the occurrence of death
Time Frame: from the beginning of study drug administration up to 18 months
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Caelyx Intravenous
Number analyzed (Participants) | 58
days | 346.0 [272.3 to 419.7]

5. Primary Outcome: Number of Participants With Partial Response
Description: Required 50 percent or greater decrease in sum of products of all bidimensionally measurable lesions without progression of assessable disease and no new lesions as measured by chest x-ray, computed tomography scan, and magnetic resonance imaging.
Time Frame: 4 weeks after chemotherapy completed
Measure: Number; unit: Participants
Arm/Group | Caelyx Intravenous
Number analyzed (Participants) | 58
Participants | 5

6. Primary Outcome: Number of Participants With Stabilization
Description: All other subjects (except complete or partial responders and those with progression [see prior definitions]) were classified as stable disease as measured by chest x-ray, computed tomography scan, and magnetic resonance imaging.
Time Frame: 4 weeks after chemotherapy completed
Measure: Number; unit: Participants
Arm/Group | Caelyx Intravenous
Number analyzed (Participants) | 58
Participants | 10

7. Primary Outcome: Number of Participants With Progression
Description: Progressive disease was defined as 25% or greater increase in the size of measurable lesion. The reappearance of any lesion or clear worsening of assessable disease or the appearance of any new lesion was also considered as progressive disease as measured by chest x-ray, computed tomography scan, and magnetic resonance imaging.
Time Frame: 4 weeks after chemotherapy completed
Measure: Number; unit: Participants
Arm/Group | Caelyx Intravenous
Number analyzed (Participants) | 58
Participants | 6

ADVERSE EVENTS:
Arm/Group | Caelyx Intravenous
Serious Adverse Events (participants affected / at risk) | 8/58
Other Adverse Events (participants affected / at risk) | 47/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caelyx Intravenous (N=58)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
ALLERGIC TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 3 (3)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
VENOUS THROMBOSIS (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caelyx Intravenous (N=58)
ANAEMIA (Blood and lymphatic system disorders) | 4 (5)
LEUKOPENIA (Blood and lymphatic system disorders) | 3 (4)
NEUTROPENIA (Blood and lymphatic system disorders) | 15 (38)
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 (4)
DIARRHOEA (Gastrointestinal disorders) | 11 (16)
FLATULENCE (Gastrointestinal disorders) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 13 (17)
STOMATITIS (Gastrointestinal disorders) | 34 (96)
VOMITING (Gastrointestinal disorders) | 4 (4)
ASTHENIA (General disorders) | 3 (3)
FATIGUE (General disorders) | 27 (45)
PYREXIA (General disorders) | 3 (5)
BODY TEMPERATURE INCREASED (Investigations) | 5 (5)
HYPOAESTHESIA (Nervous system disorders) | 3 (5)
DRY SKIN (Skin and subcutaneous tissue disorders) | 6 (9)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 4 (4)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 33 (92)
RASH (Skin and subcutaneous tissue disorders) | 13 (26)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No